CLINICAL TRIAL: NCT04039074
Title: Effects of Yoga and Relaxation on Stress and Quality of Life - a Three-armed Randomized Controlled Study
Brief Title: Effects of Yoga and Relaxation on Stress and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Relax
Record Dates: First submitted 2019-07-28; First posted 2019-07-31 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Stress, Psychological
Keywords: Yoga; Meditation; Progressive muscle relaxation; Stress; Education
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Integrative Yoga (Experimental): A 12-week "Integrative Yoga" intervention which has meditative and psycho-educational components corresponding to traditional yoga practice.
  Interventions: Behavioral: Integrative Yoga
- Iyengar yoga (Active Comparator): A 12-week established, predominantly body-oriented yoga intervention (Iyengar yoga).
  Interventions: Behavioral: Iyengar Yoga
- Mindfulness (Active Comparator): A 12-week mindfulness intervention designed for the healthy handling of stress.
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Integrative Yoga — A 12-week "Integrative Yoga" intervention which has meditative and psycho-educational components corresponding to traditional yoga practice.
  Arms: Integrative Yoga
Behavioral: Iyengar Yoga — A 12-week established, predominantly body-oriented yoga intervention (Iyengar yoga).
  Arms: Iyengar yoga
Behavioral: Mindfulness — A 12-week mindfulness intervention designed for the healthy handling of stress.
  Arms: Mindfulness

SUMMARY:
The aim of this study is to measure the effects of three stress reduction methods on patients with stress and stress associated complaints.

ELIGIBILITY:
Inclusion Criteria:

- stress with at least 4 of 10 points on the Numeric Analogue Scale (NAS) at least 1 month and at least 3 of the following 8 stress symptoms: sleep disorder, inappetence or increased appetite, shoulder neck tension/back pain, tension headache, concentration disorder, exhaustion, nervousness/irritability, stress-associated digestive problems

Exclusion Criteria:

* serious acute or chronic diseases
* pregnancy or lactation
* known serious mental illness
* immobility or restriction for gymnastics exercises due to orthopaedic, neurological or other medical cause
* participation in another study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Stress questionnaire (Cohen Perceived Stress Scale, CPSS) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Change from Baseline in the CPSS, range from 0 to 4 in each item. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the positively stated items and then summing across all scale items while higher values meaning a higher grade of perceived stress.

SECONDARY OUTCOMES:
Medical Outcomes Study Short Form Quality of Life (MOS SF-36) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-100, higher score meaning a better outcome
Hospital Anxiety and Depression Scale (HADS) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-42, lower score meaning a better outcome
Zerssen symptom list (B-LR and B-LR') | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 20-80, higher score meaning a better outcome
International Physical Activity Questionnaire (IPAQ) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  MET minutes represent the amount of energy expended carrying out physical activity. To get a continuous variable score from the IPAQ (MET minutes a week) we will consider walking to be 3.3 METS, moderate physical activity to be 4 METS and vigorous physical activity to be 8 METS.
Maslach Burnout Inventory (MBI) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-96, higher score meaning a better outcome
Mindfulness (Freiburger Fragebogen zur Achtsamkeit, FFA) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-56, higher score meaning a better outcome
Aspects of Spirituality (ASP) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-112, higher score meaning a better outcome
Self-Regulation | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 16-96, higher score meaning a better outcome
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-160, higher score meaning a better outcome
Trauma symptoms (Posttraumatic Checklist, PCL-5) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-80, higher score meaning a better outcome
Mysticism Scale Short Form | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing full scale, range 0-32, higher score meaning a better outcome
Numerical Analog Scales | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Assessing stress, back pain, headache, shoulder/neck tension, sleep quality, exhaustion, nervousness, digestive complaints, mood on 0-11 points each.
Expectation questions | Date of inclusion (baseline)
  For intervention 1, intervention 2 and intervention 3 on a 6-point likert scale from 1 (very strong) to 6 (nothing at all)
Evaluation questions | After 12 weeks, after 24 weeks
  For intervention 1, intervention 2 and intervention 3 on a 6-point likert scale from 1 (very strong) to 6 (nothing at all)
Bio-electrical Impedance Analysis (BIA) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Estimation of the body composition via bio-electrical impedance analysis (muscle mass in kg)
Dietary Behaviour assessed by Food Frequency Questionaire (Gesundheit Erwachsener in Deutschland, DEGS) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Quantitative description of nutritional habits
Medication intake | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Name of medication and dosage
Heart Rate Variability (HRV) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  24h measuring by Faros 180 (chest)
Sociodemographic Measurements | Date of inclusion (baseline)
  Age, gender, education level, household income, employment status, marital status, language spoken, complete family history, current and previous illness and co-morbidities, and current medications
Behavioral questions: alcohol consumption | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Number of alcoholic beverages on average per week in the last month
Behavioral questions: relaxation | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Relaxation behavior on average per week in the last month in minutes
Behavioral questions: cigarettes | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  Number of cigarettes on average per week in the last month in minutes
Electrodermal Activity (Galvanic Skin Response) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  24h measuring by Biovotion Everion device
Blood Volume Pulse | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  24h measuring by Biovotion Everion device
Respiration Rate | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  24h measuring by Biovotion Everion device
Interbeat Interval (IBI) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  24h measuring by Biovotion Everion device
Heart Rate (HR) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  24h measuring by Faros 180 (chest), Biovotion Everion
Skin Temperature | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  24h measuring by Biovotion Everion device
Blood Oxygenization | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  24h measuring by Biovotion Everion device
Body weight (kg) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
  24h measuring by Biovotion Everion device
Body Mass Index (kg/m2) | Date of inclusion (baseline), after 12 weeks, after 24 weeks
Waist circumference (cm) | Date of inclusion (baseline), after 12 weeks, after 24 weeks

OTHER OUTCOMES:
Qualitative interviews in focus groups interviews | 12 weeks after inclusion
  Qualitative assessment will be carried out in 45-minute focus group interviews in 12 (randomized selected) patients participating in the study. The interviews will be recorded, transcribed and analyzed with qualitative content analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite - Universitätsmedizin Berlin
Locations (1):
- Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes